CLINICAL TRIAL: NCT07315399
Title: The Correlation Between Obstructive Sleep Apnea-Related Nocturnal Hypoxemia Parameters and Coronary Microvascular Dysfunction: A Prospective Cohort Study
Brief Title: The Correlation Between Obstructive Sleep Apnea-Related Nocturnal Hypoxemia Parameters and Coronary Microvascular Dysfunction: A Prospective Cohort Study (SLEEP-CMD)
Acronym: SLEEP-CMD
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingAnzhen
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: OSA - Obstructive Sleep Apnea; Coronary Microvascular Dysfunction (CMD); Coronary Artery Disease (CAD)
Keywords: OSA - Obstructive Sleep Apnea; Coronary Microvascular Dysfunction; Coronary Artery Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Coronary Artery Disease | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography — 1. Polysomnography (PSG) All patients underwent overnight polysomnography using a diagnostic system during their hospitalization. The following nocturnal respiratory parameters were recorded: Apnea-Hypopnea Index (AHI), heart rate-related parameters (MaxHR, MHR, MinHR), Oxygen Desaturation Index (ODI), mean apnea duration, longest apnea duration, mean hypopnea duration, longest hypopnea duration, minimum oxygen saturation (minSpO2), and the percentage of time with oxygen saturation below 90% (T90).
  2. Angio-IMR Assessment Data Acquisition and Technique: Clear angiographic images of the LAD, LCX, and RCA were acquired from at least two different projection angles. Images were required to be free of vessel overlap and foreshortening. Three-dimensional reconstruction and hemodynamic calculations were performed using dedicated software (AccuIMR, Version 1.0; ArteryFlow Technology, Hangzhou, Zhejiang, China).An Angio-IMR value > 25 U was defined as the threshold for diagnosing CMD.
  Other Names: Angiography-derived Index of Microvascular Resistance

SUMMARY:
In a cohort of patients with suspected myocardial ischemia undergoing sleep studies, the objectives of this study were:

1. To determine the association between various obstructive sleep apnea (OSA)-related nocturnal hypoxemia parameters and coronary microvascular dysfunction (CMD) in patients with suspected myocardial ischemia.
2. To compare the predictive value of nocturnal hypoxemia parameters versus the traditional Apnea-Hypopnea Index (AHI) for coronary microvascular dysfunction.
3. To evaluate the prognostic value of nocturnal hypoxemia parameters in predicting Major Adverse Cardiovascular Events (MACE) during the follow-up period.
4. To explore the potential mediating roles of inflammatory and oxidative stress biomarkers in the relationship between nocturnal hypoxemia parameters and coronary microvascular dysfunction.

DETAILED DESCRIPTION:
Coronary Microvascular Dysfunction (CMD) constitutes the core pathological mechanism underlying Ischemia with Non-Obstructive Coronary Arteries (INOCA) and serves as a significant etiological factor in Ischemic Heart Disease (IHD). CMD exhibits a high prevalence within the cardiovascular disease population and is significantly associated with the risk of Major Adverse Cardiovascular Events (MACE). A meta-analysis has demonstrated that all-cause mortality in patients with CMD is 3.93 times higher than in the non-CMD population, with a 5.16-fold increase in the risk of MACE. Obstructive Sleep Apnea (OSA) is a highly prevalent sleep-disordered breathing condition, affecting approximately 936 million people globally and 176 million adults in China. As a critical cardiovascular comorbidity, OSA has a detection rate as high as 50%-83% among patients with Cardiovascular Disease (CVD) and is closely related to the development and progression of heart failure and atrial fibrillation. OSA can significantly promote the onset and progression of CMD through intermittent hypoxia-induced oxidative stress, the release of pro-inflammatory cytokines, and enhanced sympathetic nervous activity. Therefore, exploring the interaction mechanisms between CMD and OSA holds significant clinical value.

The core pathological features of CMD involve structural remodeling and functional abnormalities of the coronary microvasculature. The gold standard for its diagnosis is the Index of Microvascular Resistance (IMR) measured via an invasive pressure wire; however, this procedure is complex. In contrast, the Angiography-derived Index of Microvascular Resistance (Angio-IMR) is simple to perform, and numerous clinical studies have confirmed its high consistency with invasive IMR. Currently, an Angio-IMR >25 U is considered the cutoff value for diagnosing CMD. The typical clinical presentation of OSA includes habitual snoring, morning fatigue, excessive daytime sleepiness, and sleep fragmentation. Its diagnosis relies on Polysomnography (PSG), and disease severity is quantified and graded using the Apnea-Hypopnea Index (AHI).

Previous studies have confirmed an independent correlation between OSA and CMD; however, existing evidence is largely based on single assessments using the AHI, lacking a systematic analysis of hypoxemia characteristics. While AHI reflects the overall frequency of respiratory events, it cannot effectively distinguish the severity, duration of exposure, and frequency of hypoxemia. Existing evidence suggests that at identical AHI levels, the 5-year incidence of cardiovascular events can differ by up to 2.3-fold among patients with different hypoxia patterns. Furthermore, intervention strategies based solely on AHI have shown limited efficacy in improving all-cause mortality in CVD patients with comorbid OSA. Our team's preliminary retrospective cohort study indicated that the minimum oxygen saturation (minSpO2) ≤90% and the time with oxygen saturation below 90% (T90) were independently associated with CMD, whereas no significant correlation was found between AHI and CMD. This suggests that nocturnal hypoxemia parameters may offer superior predictive value for OSA-related CMD risk compared to the traditional AHI metric. However, clear evidence regarding the dose-response relationship between hypoxic parameters and CMD is currently lacking, and the specific impact of different hypoxic patterns (intermittent vs. sustained hypoxia) on the pathogenesis of CMD remains unelucidated. This limits the precise risk stratification and the formulation of individualized intervention strategies for CMD in OSA patients. Therefore, this study proposes a prospective cohort study to systematically evaluate the association and mechanisms between OSA-related nocturnal hypoxemia parameters and CMD. The aim is to construct a cardiovascular risk stratification model for OSA patients based on hypoxic characteristics, providing a scientific basis for implementing personalized targeted interventions, and ultimately improving patients' clinical prognosis and health-related quality of life.

The current study will be conducted by the National clinical research center for cardiovascular disease at multiple collaborating centers across China.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years, of any gender.
2. Scheduled for elective coronary angiography due to symptoms or evidence of myocardial ischemia.
3. Agreed to and capable of completing overnight polysomnography (PSG) monitoring.
4. Provided written informed consent and were willing and able to comply with baseline assessments and long-term follow-up.

Exclusion Criteria:

1. Presence of coronary chronic total occlusion (CTO), history of coronary artery bypass grafting (CABG), severe valvular heart disease, dilated or hypertrophic cardiomyopathy, congenital heart disease, or heart failure (NYHA functional class III-IV).
2. Sleep-disordered breathing with central sleep apnea (CSA) as the primary manifestation.
3. Severe hepatic insufficiency (Child-Pugh class C) or renal failure (eGFR < 30 mL/min/1.73 m²).
4. Pregnancy or lactation.
5. Life expectancy of less than 2 years, or any other condition that the investigators considered unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected myocardial ischemia patients underwent PSG to acquire detailed parameters of OSA-related nocturnal hypoxemia.
Sampling Method: Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
the Prevalence of CMD Among Patients with OSA of Different Severities | at 6, 12, and 24 months after discharge
  Differences in the Prevalence of Coronary Microvascular Dysfunction Among Patients with Obstructive Sleep Apnea of Different Severities

SECONDARY OUTCOMES:
The composite endpoint of major adverse cardiovascular events (MACE) | At 6, 12, and 24 months after discharge
  including cardiac death, non-fatal myocardial infarction, and rehospitalization for unstable angina or heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Due to patient privacy and ethical restrictions.

REFERENCES:
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439